CLINICAL TRIAL: NCT07407153
Title: Ultrasound Based Triaging of Women With Breast Lump on Clinical Breast Examination: A Pilot Study, Indonesia, 2025-28
Brief Title: Triaging of Women Detected With a Breast Lump on Clinical Breast Examination Using Portable Ultrasound Device
Acronym: Ultra-3 CBE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Dharmais National Cancer Center Hospital (Other Government)
Responsible Party: Principal Investigator, Ravivarman Lakshmanasamy, Public Heatlh Officer, International Agency for Research on Cancer
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IARC IEC 25-12
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: breast; breast carcinoma; triage; ultrasound; portable device
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All women detected with a breast lump on clinical breast examination, who have consented for study (Experimental): The identified women will be subject to ultrasound triaging, and those with non-cystic lesions will be referred for further evaluation
  Interventions: Diagnostic Test: Portable ultrasound device

INTERVENTIONS:
Diagnostic Test: Portable ultrasound device — The women detected with a breast lump on clinical breast examination will be examined using a portable ultrasound device by a trained medical officer at the primary healthcare facility, to traige them

SUMMARY:
This study aims to stratify women diagnosed with a lump in the breast by clinical breast examination(CBE) using a hand-held ultrasound machine. They will be stratified either with benign or potentially malignant lesion. As most of the lesions identified by CBE are benign, stratifying them (triage) avoids the unnecessary procedures in terms of mammography and biopsy. This will also reduce the burden in the further assessment sites, and provide better quality services in these places.

DETAILED DESCRIPTION:
The project nested in the national breast cancer screening programme of Indonesia aims to determine whether ultrasound-based triaging by trained medical officers at primary health facilities can detect benign lesions in women with breast lumps identified through clinical breast examination (CBE) at these facilities. This point-of-care approach would help reduce the load on tertiary facilities at radiology and pathology centers and also prevent unnecessary interventions in women diagnosed with benign breast lesions in a CBE-based screening programme.

Primary Objective

* To determine the positive and negative predictive value of clinical breast examination in detecting malignancies when ultrasound-based triaging is performed by trained medical officers on women found positive through clinical breast examination Secondary objectives
* To determine the sensitivity and specificity of ultrasound-based triaging by trained medical officers at primary health centres by excluding the benign masses in breast
* To assess the outcomes of ultrasound-based triaging through early follow up screening of the women excluded from undergoing further evaluation
* To assess the feasibility and acceptability of taking up ultrasound-based triaging by trained medical officers at primary health centres as part of routine breast cancer screening pathway

Methods:

Study design:

A prospective study will be conducted among the women attending breast cancer screening clinics in selected five primary health facilities in West Jakarta, Indonesia. As a pre-requisite, the medical officers in the primary health facilities will be trained by radiologists from the Dharmais hospital in performing basic ultrasound techniques to identify benign (cysts/fibrocystic disease) lesions in the breast. A benign lesion will be defined as an oval or round, circumscribed, hypoechoic lesion in parallel orientation with no posterior features in the ultrasound finding. Additional information on the characteristics of a benign breast lesion in ultrasound imaging is available in the IARC platform.

Study Procedure:

We will recruit women (aged 30 to 69 years) who undergo clinical breast examination and are found to be detected positive with a lesion in the breast at the identified PHCs. The participating women will be explained about the study and a written informed consent will be obtained. The participants will then be interviewed by trained female health worker/nurse to collect the socio-demographic and reproductive health related data in conﬁdential settings.

The trained medical officers will perform the ultrasound examination of the breast identified with lesions in breast by clinical breast examinations. The probe will be applied to the area suspected to be abnormal on CBE to detect the purely cystic lesions in the breast. Women with pure cystic lesions or no abnormalities detected on ultrasound will be reassured. However, it will be explained to them that ultrasound cannot completely rule out a breast cancer. Hence, they will be advised to undergo repeat CBE examination after one year. Additionally, a subset (20%) of women who are detected with non-malignant lesions or no lesions based on ultrasound-based triaging will be selected at random and sent to Dharmais Hospital for further evaluation. This will enable address the verification bias component also.

The remaining set of women with potential malignant lesions will be referred for further diagnostic workup at the Dharmais tertiary care hospital.

Study period:

The study period is till February 2028, with 24 months for recruitment of adequate number of sample size with additional months for follow up of the set of women who were excluded from diagnostic work up following identification of the lesion to be benign by ultrasound examination.

Study population:

Women undergoing the clinical breast examination within the target age and found with a lesion in breast will be considered to be included for the study after they provide written informed consent.

Non-inclusion criteria:

* Women already screened in the last three years
* Women with known history of breast cancer or breast surgery
* Symptomatic with high probability of breast cancer diagnosis (ulcerated lump, blood-stained nipple discharge etc.)
* Debilitating illness
* Unable to provide informed consent due to certain mental illnesses
* Unlikely to be compliant to study procedures and/or follow up as determined by the investigator Sample size

The sample size has been calculated using invasive breast cancers as the outcome of interest. In order to demonstrate that use of ultrasonography can lead to an increase in PPV after screening with CBE, we used the following assumptions:

* A 5% PPV of CBE to detect breast cancers
* A 50% relative increase in PPV if ultrasonography triage is used for abnormal after screening with CBE
* A total loss to follow-up of 10%;
* A 80% power; and
* A 5% level of significance.

The total sample size of 598 women abnormal on CBE will be required. A secondary data analysis of the national cancer screening data by the National NCD division of Indonesia mentions that 5.4% of the screened target population was detected with breast mass.

Considering the age group (30 to 69) in this study, to identify around 600 women positive on CBE, around 10,000 women in the target age group have to screened by CBE.

ELIGIBILITY:
Inclusion Criteria:

* Women eligible for breast cancer screening as per the National screening programme in the country, and those detected with a breast lump on clinical breast examination

Exclusion Criteria:

* Women already screened in the last three years
* Women with known history of breast cancer or breast surgery
* Symptomatic with high probability of breast cancer diagnosis (ulcerated lump, blood-stained nipple discharge etc.)
* Debilitating illness
* Unable to provide informed consent due to certain mental illnesses
* Unlikely to be compliant to study procedures and/or follow up as determined by the investigator

Ages: 30 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women eligible for breast cancer screening in the study site country
Enrollment: 600 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value and negative predictive value of CBE by ultrasound triaging | From recruitment to 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dharmais hospital, Jakarta, West Jakarta, Indonesia